CLINICAL TRIAL: NCT04886310
Title: Turkish Validity and Reliability Study of Peabody Developmental Motor Scale-2 in Infants Aged 0 - 24 Months
Brief Title: Peabody Developmental Motor Scale-2 in 0 - 24 Months in Turkey
Status: Completed | Type: Observational
Sponsor: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Nilay Comuk Balci, Pt, PhD, Associate Professor, Ondokuz Mayıs University
Other Study IDs: 41901325-050.99
Record Dates: First submitted 2021-05-10; First posted 2021-05-14 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Motor Development; Infant, Premature, Diseases
Keywords: validity; Peabody Developmental Motor Scale II (PDMS-2); motor development
MeSH Terms: conditions — Infant, Premature, Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Peabody Developmental Motor Scale II (PDMS-2) — is composed of six subtests (reflex, stationary, locomotion, object manipulation, grasping, and visual-motor integration) that measure inter-related abilities in early motor development. It was designed to assess gross and fine motor skills in children from birth through 5 years of age.

SUMMARY:
This study is the determination of the Turkish version of the Peabody Developmental Motor Scale-2 and its Turkish validity reliability in infants age between 0 - 24 months and to spread its use for evaluation in early rehabilitation in our country.

DETAILED DESCRIPTION:
There are developments in the field of diagnosing children with a high risk of developmental disorders such as cerebral palsy (CP), mental problems and autism spectrum disorder in infancy . In particular, in infants experiencing the onset of extrauterine life in the neonatal intensive care unit, the combination of neonatal neuroimaging along with the assessment of general movements results in a highly accurate prediction of CP .A clinical tool often used in predictions is a neurological examination. Various standard variants are available, such as the Hammersmith Infant Neurological Examination (HINE), Alberta Infant Motor Scale (AIMS). PGMS-2 was developed by Folio and Fewell (2000) to determine the gross and fine motor development levels of children from birth to 71 months. The scale can be used for both children with healthy development and children with special needs. In the development of the Peabody Developmental Motor Scale (PGMS), which is the original version of PGMS-2 used in this study, a developmental structure was adopted instead of sticking to a certain theoretical perspective. PGMS is the first nationally standardized assessment tool that gives gross and fine motor scores separately in the United States of America (USA).This study is the determination of the Turkish version of the Peabody Developmental Motor Scale-2 and its Turkish validity reliability in infants age between 0 - 24 months and to spread its use for evaluation in early rehabilitation in our country.

ELIGIBILITY:
Inclusion Criteria:

* Infants between 0-24 months (adjusted age for premature infants will be calculated),who are followed as neurologically and developmentally at risk infants
* Infants who are not in neonatal intensive care unit

Exclusion Criteria:

* Infants with congenital heart problems
* Infants of families who do not accept the study
* Infants with musculoskeletal system anomaly
* Infants connected to respiratory equipment

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Infants between 0-24 months (adjusted age for premature infants will be calculated),who are followed as neurologically and developmentally at risk infants
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2020-09-10 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Peabody Developmental Motor Scale II (PDMS-2) | 45-60 minutes
  is composed of six subtests (reflex, stationary, locomotion, object manipulation, grasping, and visual-motor integration) that measure inter-related abilities in early motor development. It was designed to assess gross and fine motor skills in children from birth through 5 years of age.

SECONDARY OUTCOMES:
The Alberta Infant Motor Scale (AIMS) | 30-40 minutes
  The AIMS is a norm-referenced observational scale that enables the determination of infants with delay or deviation in motor development and to evaluate the changes in motor development over time. It is used to follow the movement patterns of infants who show atypical movement patterns over time. Average application time is 30-40 minutes. 0-18. The evaluation is made on a total of 58 items in 4 different developmental positions: supine, prone, sitting and standing between months.
Hammersmith Infant Neurological Examination (HINE) | 30-45 minutes
  The HINE includes three sections, the Neurological Examination, the Development of Motor Functions and the State of Behaviour. The first section evaluates cranial nerve, posture, movements, tone and reflexes. These items are not age-dependent. The second section evaluates head control, sitting, voluntary grasping, rolling, crawling and walking. The third section evaluates state of consciousness, emotional state and social orientation.

CONTACTS AND LOCATIONS:
Overall Officials: NILAY ÇÖMÜK BALCI, Pt,PhD, Principal Investigator — Ondokuz Mayıs University
Locations (1):
- Nilay Çömük Balci, Samsun, Atakum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided